CLINICAL TRIAL: NCT00453167
Title: A Phase II Study of Weekly Paclitaxel and Gemcitabine as Second-line Therapy in Patients With Metastatic or Recurrence Small Cell Lung Cancer
Brief Title: Weekly Paclitaxel Plus Gemcitabine as Second-line in Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Heung Tae Kim, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-155
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
Keywords: Small cell lung cancer; second-line therapy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80mg/m2 iv on day 1 and 8, every 3 weeks until disease progression
Drug: Gemcitabine — Gemcitabine 1000mg/m2 iv on day 1 and 8, every 3 weeks until disease progression

SUMMARY:
As a single agent, paclitaxel has a response rate of 33% and 25-29% in SCLC patients with sensitive relapse and with resistant relapse, respectively. As a single agent, gemcitabine also has a response rate 16% and 6-13% in SCLC patients with sensitive relapse and with resistant relapse, respectively. Because of single-agent activity, different mechanism of action, non-overlapping toxicities, and beneficial pharmacologic interaction, paclitaxel and gemcitabine combinations are attractive for testing in clinical trials.

DETAILED DESCRIPTION:
The treatment consists of paclitaxel 80 mg/m2 and gemcitabine 1,000 mg/m2 given intravenously on days 1 and 8 of a 21-day cycle.

Patients receive treatment every 3 weeks till disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed SCLC
2. Clinically diagnosed metastatic or recurrent SCLC according to Sixth Edition of the AJCC Cancer Staging Manual
3. At least 18 years old
4. ECOG performance status 0-2
5. Disease status must be that of measurable disease defined as RECIST:Lesions that can be accurately measured in at least one dimension > 10 mm with chest x-ray, spiral CT scan or physical examination
6. Progression during or after prior first line chemotherapy or chemoradiotherapy.
7. Before study entry, a minimum of 21 days must have elapsed since any prior chemotherapy or radiation
8. No prior radiotherapy to measurable lesion(s) but previous surgery and/or chest radiotherapy for the primary lesion is allowed
9. Adequate major organ function including the following:Hematologic function: WBC ≥ 3,500/mm3 or absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥ 100,000/mm3Hepatic function: bilirubin ≤ 1.5 x UNL , AST/ALT levels ≤ 2.5 x UNLRenal function: serum creatinine ≤ 1.5mg/dL
10. Patients should sign an informed consent
11. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study registration.

Exclusion Criteria:

1. MI within preceding 6 months or symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmia
2. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complication of study therapy
3. Other malignancy with the past 5 years except adequately treated cutaneous basal cell carcinoma or uterine cervix in situ cancer
4. Pregnant or nursing women
5. Psychiatric disorder that would preclude compliance.
6. Major surgery other than biopsy within the past two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-12; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate of paclitaxel plus gemcitabine | the ratio between the number of responders and number of patients assessable for tumor response

SECONDARY OUTCOMES:
To access the toxicity | the first day of the treatment to 30 days after the last dose of study drug
To estimate the time to progression | the first day of treatment to the date that disease progression is reported
To examine the association between genotypes of paclitaxel biotransformation and the pharmacokinetics / | before the first treatment date, each response evaluation until disease progression
To estimate the overall survival | the first day of treatment to death date

CONTACTS AND LOCATIONS:
Overall Officials: Heung Tae Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea